CLINICAL TRIAL: NCT02723292
Title: City of Rochester Teen Outreach Program (TOP™) Evaluation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: State University of New York at Binghamton, Decker School of Nursing (Unknown); City of Rochester Department of Recreation and Youth Services (Unknown)
Responsible Party: Principal Investigator, Hugh Crean, Assistant Professor, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 36508
Record Dates: First submitted 2016-02-04; First posted 2016-03-30 (Estimated); Last update posted 2018-02-12 (Actual); Status verified 2018-02

CONDITIONS: Adolescent Problems; Sex Behavior; Academic Underachievement Disorder of Childhood or Adolescence
MeSH Terms: conditions — Sexual Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental group services (Experimental): This study will replicate the evidence-based TOP™ in after-school sessions held during RC hours. The primary components of TOP™ include: Comprehensive age-appropriate sexuality education; 90-minute sessions, once a week after-school, during the school year for nine months, using the Changing Scenes© curriculum, and at least twenty hours of youth-led service learning, which involves youth in planning, implementing and reflecting on, community service and leadership.
  Interventions: Behavioral: TOP
- Control group services (Active Comparator): Youth in the control arm will receive a work readiness training curriculum focused on competencies to secure employment. This will include such topics as building customer service skills, clear and direct communication, and creating a work portfolio.
  Interventions: Behavioral: Control intervention

INTERVENTIONS:
Behavioral: TOP
  Arms: Experimental group services
Behavioral: Control intervention
  Arms: Control group services

SUMMARY:
As part of a 5-year national effort to reduce teen pregnancy, the University of Rochester is partnering with the City of Rochester Department of Recreation and Youth Services to evaluate the City's replication of the Teen Outreach Program (TOP™) for 11-14 year old youth registered at 11 selected Recreation Centers (RCs). A youth development program with demonstrated efficacy to reduce teen pregnancy, school failure and drop-out rates, TOP™ has never been studied in RCs. Advancing from efficacy to effectiveness, the investigators will also measure program fidelity obtained in RCs.

ELIGIBILITY:
Inclusion Criteria:

* must be registered at a participating RC
* age 11 through 14 years
* participants must assent and parent(s) or legal guardian(s) provide permission to participate
* basic understanding of the English language

Exclusion Criteria:

* age at enrollment of less than 11 or greater than 14 years
* for facilitators, age less than 21 is an exclusion criterion

Ages: 11 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1188 (Actual)
Dates: Start 2011-09; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Number of participants who become pregnant | 21 months
Number of youth who report ever having had sexual intercourse | 21 months
  For youth who were sexually naive at baseline, the outcome is the number of youth who report ever having had sexual intercourse at the 21 month assessment point.
Amount of sexual intercourse in preceding 3 months without an effective means of birth control | 21 months
  The number of times a youth reports having had sexual intercourse without using an effective means of birth control measured at the 21 month assessment point.

SECONDARY OUTCOMES:
Number of failing grades on report card | 21 months
  This is a self-report measure of the number of courses failed on the last report card received, measured at the 21 month assessment point.

IPD SHARING:
Plan to Share IPD: Undecided